CLINICAL TRIAL: NCT00292318
Title: Biofeedback Therapy for Fecal Incontinence a Randomized Control Trial
Brief Title: Treatment of Patients With Fecal Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue due to medical equipment necessary for research study was removed from facility.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-013-05S
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Fecal Incontinence
Keywords: adequate relief; anorectal manometry; biofeedback therapy; fecal incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Control group of patients with fecal incontinence which would be given medical therapy and exercises to perform as treatment.
  Interventions: Behavioral: control group
- Arm 2 (Experimental): Study group of patients with fecal incontinence which would be given biofeedback therapy and exercises to perform as treatment.
  Interventions: Behavioral: Biofeedback Therapy for Fecal Incontinence: A Randomized Control Study

INTERVENTIONS:
Behavioral: Biofeedback Therapy for Fecal Incontinence: A Randomized Control Study — Patients who have more than one episode per week of fecal incontinence would be enrolled and randomized into either the control group (medical counseling and exercises) or study group (biofeedback therapy, medical counseling, and sphincter exercises) for seven sessions to assist with their medical problem.
  Arms: Arm 2
Behavioral: control group — Medical counseling and ano-sphinctal exercises.
  Arms: Arm 1

SUMMARY:
The purpose of this study is to determine if a behavioral treatment method called biofeedback will reduce the frequency of episodes of leakage of fecal material in patient suffering from fecal incontinence.

DETAILED DESCRIPTION:
Fecal incontinence (FI) is a devastating condition that causes psychological stress, shame, embarrassment, and social isolation. It has a major impact on quality of life of patients and their families. It complicates medical illnesses and management, has major economic consequences and can contribute to early nursing home placement. Although FI affects 2.2% to 11% of the general population, the magnitude of the problem is underestimated, since most patients do not discuss this silent affliction with their care providers. In uncontrolled studies of biofeedback for FI, including our preliminary observations in male veterans without anal sphincter injury, improvement was observed in up to 80% of patients. However, it may not be appropriate for all patients. One recent randomized, controlled trial in predominantly (93% women) female patients, many (> 60%) with post-obstetrical anal sphincter injury, reports that biofeedback is no more effective than medical therapy alone. The trial provides data for the formulation of an evidence-based approach to treat FI in female veterans. There are no randomized, controlled data on the effectiveness of biofeedback for FI in male patients. A randomized, controlled trial is needed to assess the effectiveness of multi-component biofeedback therapy versus standard medical therapy in man. The immediate objectives of the current proposal are to evaluate the effectiveness of biofeedback treatment for FI and to identify baseline patient characteristics that will predict improvement and adequate relief in FI symptoms following treatment. This will lead directly to our long-term goal of providing optimal treatment for FI by tailoring biofeedback plus medical therapy to each patient's needs, based on sound clinical evidence. This project is a prospective, randomized, controlled clinical trial comparing two treatments for FI among patients who have failed medical treatment under the care of their primary care providers and are referred for evaluation and management of current FI. As part of standard care, all referred patients will receive a history and physical examination, including medical, surgical, FI-specific symptoms and physical findings (general, mobility, mental status and anorectal examination). Those who meet inclusion criteria and who agree to participate will be randomly assigned to one of 2 study arms: 1. medical therapy alone, 2. medical therapy + sphincter strength + sensation + coordination training. Baseline data will also include adequate relief measure, incontinence scores based on bowel habit diary, anorectal parameters based on manometric and sensory testing, general and FI-specific quality of life, depression, anxiety, and expectation of improvement following treatment. All questionnaires will be based on published, validated instruments. Patients will be treated in six biweekly sessions (3 months). Medical therapy (six 40 - 60 minute sessions) includes advice, medication for constipation/diarrhea, and instruction related to empiric anal sphincter exercises (group 1). Biofeedback treatment (six 40 - 60 minute sessions) includes medical therapy plus all components of biofeedback (groups 2). Follow up data will be obtained in all patients at the end of treatment (3 months) and by mailed questionnaires at 12 months after completion of treatment or dropout. We can determine if biofeedback plus medical therapy will be superior to medical therapy alone in providing FI symptom relief. The possibility that more patients will report relief of FI symptoms when specific deficit(s) detected at baseline testing show(s) improvement with treatment. The influence of co-variables on results of treatment can also be determined. Our long term goal is to develop a clinically relevant strategy that will be cost-effect for the management of FI in VA patients (predominantly male) within the organizational frame work of primary and subspecialty care. If biofeedback treatment is proven to be effective, and VA patients can be offered therapy components with optimal likelihood of success, the obvious benefit to our VA patients is abatement of the silent affliction of FI and improvement in patient satisfaction and quality of life. Further study will focus on a multi-site cooperative study to assess which component of biofeedback is most instrumental in bringing about improvement and relief in patients with specific deficits.

ELIGIBILITY:
Inclusion Criteria:

Male or female patient with inadequate relief of fecal incontinence symptoms after documented management in the primary care setting. They must have:

* a mini-mental status score of > 18
* an "up and go" test score of < 30 seconds
* bowel habit diary showing > one episode of fecal incontinence episode per week

Exclusion Criteria:

* patients who previously underwent a course of biofeedback for fecal incontinence
* age < 18 years
* major neurological disease
* significant cognitive impairment (mini mental status examination score < 18), functional impairment (up and go score of > 30 seconds)
* active inflammatory bowel disease
* history of spinal cord injury
* rectal resection
* ileal pouch procedures
* latex allergy
* significantly distressed and unable to consider informed consent issues adequately
* needing urgent medical referral
* insufficient written English skills to complete the questionnaires
* require surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix W Leung, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

REFERENCES:
- See also: One of the family of web sites by the international Organization for Functional Gastrointestinal Disorders (IFFGD) — http://www.aboutincontinence.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control group of patients with fecal incontinence which would be given medical therapy and exercises to perform as treatment.
  control group: Medical counseling and ano-sphinctal exercises.
- Study Grp/Biofeedback: Study group of patients with fecal incontinence which would be given biofeedback therapy and exercises to perform as treatment.
  Biofeedback Therapy for Fecal Incontinence: A Randomized Control Study: Patients who have more than one episode per week of fecal incontinence would be enrolled and randomized into either the control group (medical counseling and exercises) or study group (biofeedback therapy, medical counseling, and sphincter exercises) for seven sessions to assist with their medical problem.
Period: Overall Study
Arm/Group | Control | Study Grp/Biofeedback
Started | 4 | 3
Completed | 2 | 2
Not Completed | 2 | 1
Not completed — Study terminated by officials | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Study Grp/Biofeedback | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Patient Report of "Adequate Relief" From FI Symptoms With a "Yes" Answer Will be Used as Primary Outcome Variable. Data Will be Recorded at End of Treatment. A "Responder" Will be Defined as One Who Provides a "Yes" Answer.
Description: Only reporting the results of participants who reported adequate relief.
Time Frame: The primary outcome will be determined at the end of the study which will be 20 weeks after starting the study.
Population: Only participants that completed the full number of study visits were analyzed.
Measure: Number; unit: participants
Arm/Group | Control | Study Grp/Biofeedback
Number analyzed (Participants) | 2 | 2
participants | 2 | 2

2. Secondary Outcome: Change in Anorectal Physiologic Tests (Absolute Squeeze Pressure)
Description: Measurement of pressure changes by a colonoscope as recorded by a manometric catheter connected to a Polygraph transducer.
Time Frame: The secondary outcome will be determined at the end of the study which will be 20 weeks after starting the study.
Population: Data were not collected due medical instruments to measure this outcome were removed by VA staff causing the study to be terminated.
Arm/Group | Control | Study Grp/Biofeedback
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Study Grp/Biofeedback
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes